CLINICAL TRIAL: NCT04568382
Title: The Impact of Life Context and Social Determinants of Health on Treatment Burden in Diabetes and Multiple Chronic Conditions
Brief Title: Diabetes Communication and Treatment Burden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Elizabeth Marianne Magnan, Associate Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1619593
Record Dates: First submitted 2020-09-11; First posted 2020-09-29 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2; Multiple Chronic Conditions
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Enhanced PVP
  Interventions: Other: CI-PVP (context-informed pre-visit planning)
- Standard (Active Comparator): Standard PVP
  Interventions: Other: Standard PVP (pre-visit planning)

INTERVENTIONS:
Other: CI-PVP (context-informed pre-visit planning) — may experience a single additional phone call from clinic staff in addition to the standard clinic staff chart review, email and/or phone call prior to diabetes office visit
  Arms: Intervention
Other: Standard PVP (pre-visit planning) — standard clinic staff chart review, email and/or phone call prior to diabetes office visit
  Arms: Standard

SUMMARY:
The objective of this proposal is to pilot test two types of pre-visit planning, where clinical staff reviews charts and talks to patients before their doctors appointments, to reduce the burden of diabetes care on the patient without increasing the visit workload during busy primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* patient at the UCD ACC family medicine residency clinic
* age 18+,
* has diabetes per Diabetes Registry (HealthyPlanet2020)
* PLUS at least one other chronic condition
* attends a primary care office visit (in-person or telehealth) during the study initial data collection period with a physician who is participating in the study
* speaks and writes English well enough to complete a written or oral survey
* consents to participate

PCPs:

-sees patients as a primary care physician at the study clinic site

Exclusion Criteria:

* does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pilot feasibility | at completion of study, 4 months after last study visit
  patients reached by phone for PVP call after assigned to call; # patients recruited successfully who were eligible; # questions completed on the surveys; # calls made to each patient and to patients total per # patients reached and # patients enrolled; # patients who completed all surveys; qualitative interviews will discuss challenges, barriers, and other feasability concerns to scaling this pilot trial to a definitive multi-center trial
Pilot acceptability) | after each clinic visit, within 2 weeks; at end of study
  a short survey measuring PCPs perception of the visit's difficulty, hassle and effort; qualittive interviews with patients, providers and those conducting the intervention PVP calls

SECONDARY OUTCOMES:
Treatment Burden of Diabetes Care Questionnaire (TBQ) | change from baseline to 4 months post visit
  a validated survey that measures patient self-assessment of chronic disease care burden; 13 items on a 5 point Likert scale, 13-65, higher score is worse
Patient Experience with Treatment and Self-Management (PETS) Questionnaire Medical Expenses Subsection | change from baseline to 4 months post visit
  a validated survey that measures patient's self-assessed ability to handle financial aspects of chronic disease care; 5 items on a 5 point Likert scale, 5-25, higher score is worse
Healthcare Climate Questionnaire (HCQ) | change from baseline to 4 months post visit
  a validated survey of patient experience with their healthcare; 6 items on a 7 point Likert scale, 6-42, higher score is better
Patient Self-Activation Measure (PAM-13) short form | change from baseline to 4 months post visit
  a validated measure of patient participation in their own healthcare; 13 items on a 4 point Likert scale, 13-52, higher score is better
Perceived Diabetes Self-Management Scale | change from baseline to 4 months post visit
  a validated survey on the patients perception of their ability to care for their diabetes; 8 items on a 5 point Likert scale, 8-40 higher score is worse
SF-12, Short Form 12 questions Health Survey | change from baseline to 4 months post visit
  a validated 12 question survey on patient's physical and mental health
Discussion of social determinants of health (SDH) during clinic visit, self-reported | after each clinic visit, within 2 weeks
  a single question survey, self-reporting by the participant, if SDH were discussed between the doctor and the patient during the visit
HgbA1c value | change from baseline to 4 months post visit
  change in A1c level from baseline to post-study, using values nearest to study start and end dates
Blood pressure measurement | change from baseline to 4 months post visit
  systolic and diastolic blood pressure value pre and psot study, using measures closest to study start and end date, and area-under-the-curve for blood pressure in between.
Body Mass Index | change from baseline to 4 months post visit
  Body Mass Index change from beginning of study to the end of the study, using most recent height available
Physician Job Satisfaction Scale | change from baseline to 4 months post visit
  validated survey on elements of physician job satisfaction
Maslach Burnout Inventory Human Services Survey for Medical Personnel | change from baseline to 4 months post visit
Depression symptoms | change from baseline to 4 months post visit
  change in symptom score, as measured by PHQ2 (0-6, higher is worse) or PHQ9 (0-27, higher is worse), as available, done within one month of study start and after visit by study end
Anxiety Symptoms | change from baseline to 4 months post visit
  change in symptom score, as measured by GAD2 (0-6, higher is worse) or GAD7 (0-21, higher is worse), as available, done within one month of study start and after visit by study end

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Magnan, MD, Principal Investigator — UCDavis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Plan to share anonymized or de-identified data per IRB approval to researchers at my institution.

REFERENCES:
- [Derived] Magnan E, Gosdin M, Tancredi D, Jerant A. Pilot randomized controlled trial Protocol: Life context-informed pre-visit planning to improve care plans for primary care patients with multiple chronic conditions including diabetes. J Multimorb Comorb. 2021 Dec 1;11:26335565211062387. doi: 10.1177/26335565211062387. eCollection 2021 Jan-Dec. PMID 34881189